CLINICAL TRIAL: NCT00581646
Title: Cross-Sectional Study of Psychosexual Impact of Cancer-Related Infertility in Women: Third Party Reproductive Assistance
Brief Title: Study of Psychosexual Impact of Cancer-Related Infertility in Women: Third Party Reproductive Assistance
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 06-110
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Cervical Cancer; Endometrial Cancer; Leukemia; Non-Hodgkin's Lymphoma; Uterine Cancer; Vaginal Cancer; Infertility
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Leukemia; Lymphoma, Non-Hodgkin; Uterine Neoplasms; Vaginal Neoplasms; Infertility | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: gynecologic cancer survivors
  Interventions: Behavioral: survey instrument
- 2: survivors of any type of malignancy with history of BMT/SCT
  Interventions: Behavioral: survey instrument
- 3: non-cancer infertile women awaiting third party reproduction
  Interventions: Behavioral: survey instrument

INTERVENTIONS:
Behavioral: survey instrument — Participants will be mailed or given a one time survey instrument and data will be collected either in person or by telephone. We expect the study survey to take approximately 35-45 minutes to complete. The domains assessed will include psychological functioning, reproductive knowledge, perception of third party reproduction and concerns, sexual functioning, and quality of life.

SUMMARY:
This study aims to learn about the needs and feelings of women who are infertile. Being infertile means not being able to have a child without the help of a third party. There are other options for building a family. The researchers are interested in the participants' thoughts about these options and want to learn about the experiences of infertile women due to cancer treatment as well as women who are infertile due to other causes. The researchers hope that what they learn will allow them to better care for infertile women in the future.

DETAILED DESCRIPTION:
As part of this study, you will be asked to fill out a series of questionnaires. These questions will ask about your feelings, sexual function, quality of life, and ideas about reproductive options. We will also ask some questions about you, your health, and your medical history. You can choose to answer these questions either at one of your doctor visits or over the telephone. You can decide the best way to complete this assessment.

ELIGIBILITY:
Inclusion Criteria:

Study group of gynecologic cancer survivors and BMT/SMT cancer survivors:

* History of a primary diagnosis of gynecologic cancer or history of any primary malignancy treated with BMT/SCT
* No evidence of disease for at least one year
* At least 18 years of age not greater than 49 years of age at time of study recruitment
* No other cancer history
* Have impaired fertility: lack of uterus but intact ovaries or lack of ovaries or lack of ovarian function based on the FSH determination but intact uterus
* Have not started or have not completed childbearing
* Able and willing to provide informed consent
* Ability to comprehend and complete questionnaire in English

Comparison Group of non-cancer infertile women awaiting egg (oocyte) donation:

* No cancer history
* At least 18 years of age not greater than 49 years of age at time of study recruitment
* In ovarian failure and on a waiting list for egg (oocyte) donation
* Have not started or have not completed childbearing
* Able and willing to provide informed consent
* Ability to comprehend and complete questionnaire in English

Exclusion Criteria:

* Inability to participate in an informed consent process
* Patients with a psychiatric disorder precluding response to the survey

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cervical cancer, Endometrial cancer, Leukemia, Non-Hodgkin's Lymphoma, Uterine cancer, Vaginal cancer survivors and non-cancer infertile women
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2006-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Investigate emotional, sexual functioning, reproductive concerns and QOL experience of 3 groups of infertile women: gynecologic cancer survivors, survivors of hematological malignancies, & the non-cancer infertile women awaiting 3rd party reproduction | 2 years

SECONDARY OUTCOMES:
Assess and describe the attitudes towards, knowledge of, and utilization of third party reproduction of the study participants (cancer and non-cancer infertile groups) | 2 years
Compare the main domains of depression, distress, sexual functioning and overall QOL of the gynecologic cancer survivors and survivors of a hematological malignancy with history of BMT/SCT to non-cancer infertile women awaiting third party reproduction | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Carter, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org